CLINICAL TRIAL: NCT07203443
Title: Child Cognitive-Affective Resilience Following 13-11 Event : A Pluridisciplinary Study of Intergenerational Transmission of a Traumatic Event
Acronym: CARE 13-11
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C21-80; 2022-A01409-34 (Other: ID RCB)
Record Dates: First submitted 2025-02-20; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Intergenerational Trauma
Keywords: Trauma; Offspring; Transmission; Psychology; Cognition; Physiology; Neuroimaging
MeSH Terms: conditions — Historical Trauma; Wounds and Injuries | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exposed group (Other)
  Interventions: Other: MRI; Other: Psychological assessment; Behavioral: Cognitive assessment; Other: Cortisol sample
- Unexposed group (Other)
  Interventions: Other: MRI; Other: Psychological assessment; Behavioral: Cognitive assessment; Other: Cortisol sample

INTERVENTIONS:
Other: MRI — Anatomical and functional MRI
Other: Psychological assessment — Inventories and clinical interviews
Behavioral: Cognitive assessment — Attention and memory tests
Other: Cortisol sample — Salivary test

SUMMARY:
CARE 13-11 study explores the transmission of trauma within families. Exposure to a traumatic event can have an impact on those directly exposed, but also on their family.

This transmission is both biological and behavioral, leading to adaptation that is still poorly understood. CARE 13-11 project offers a unique opportunity to bring together different disciplinary fields, from neuroscience to human and social sciences, to understand this phenomenon.

To answer these questions, the study includes directly exposed families with minor children born before the events, as well as families with no exposure to these events (the so-called "control" group).

ELIGIBILITY:
Inclusion Criteria:

Exposed group

Children

* Minor child born before November 13, 2015
* At least one parent was present at the scene of the attacks: criteria A1 (directly exposed to the event) or exposed to the event) or A2 (witnessed the event) of DSM-5
* With a good command of the French language (francophone)
* Whose parents have given written consent for their child's their child's participation
* At least one parent is covered by health insurance

Parent 1 (and Parent 3)

* Parent of child(ren) included
* Directly exposed to the attacks: present at the scene of the attacks: criteria A1 (directly exposed to the event) or to the event) or A2 (witness to the event) of the DSM-5
* Good command of the French language
* Affiliated with or benefiting from a social security scheme
* Has given written consent

Parent 2

* Parent of child(ren) included
* Not exposed but whose spouse (or ex-spouse) was directly exposed to the attacks on a declarative basis
* Have a good command of the French language
* Affiliated with a social security scheme or beneficiary of such a scheme
* Having given written consent

Uncle/aunt

* Not exposed, but has a brother or sister directly exposed to the attacks
* Have a good command of the French language
* Beneficiary of health insurance
* Having given written consent

Cousin

* Minor child born before November 13, 2015
* Whose aunt or uncle was directly exposed to the attacks
* Child with a good command of the French language
* Who has given written consent
* Whose parents with parental authority have given written consent for their child's their child's participation
* Whose parent is affiliated to a social security scheme or is a beneficiary of such a scheme

Unexposed group

Child

* Minor child born before November 13, 2015
* No relative (family or close friend) has been exposed to the attacks
* With a good command of the French language
* Whose parents have given their written consent for their child's their child's participation
* One of whose parents is affiliated to or benefits from a social security scheme

Parent 1

* Parent of child(ren) included
* No exposure to the attacks and no close relative (family or close friend) exposed to the attacks attacks
* No PTSD at the time of inclusion (PCL-5 < 33)
* Have a good command of the French language
* Affiliated with or benefiting from a social security scheme
* Having given written consent

Parent 2

* Parent of included child(ren)
* No exposure to terrorist attacks
* With a good command of the French language
* Affiliated with or benefiting from a social security scheme
* Having given written consent

Exclusion Criteria:

For all children:

* Loss of both parents following the events of November 13
* Presence of a history of severe neurological, mental or psychopathological disorders (epilepsy, head trauma with loss of consciousness of more than one hour, autism spectrum disorder, intellectual disability, schizophrenia)
* Persons subject to a legal protection measure (safeguard of justice, curatorship, guardianship)
* Subject to a period of exclusion in the context of another research project
* Refusal of the child to participate in research

For children undergoing the on-site protocol:

* Person with contraindications to MRI
* For women of childbearing age, pregnancy in progress
* Psychotropic products capable of modifying attention, vigilance and concentration taken less than 24 hours before questionnaires or examinations (sleeping pills and hypnotics, antipsychotics, mood regulators, antiepileptics and antihistamines). If in doubt about the patient's ability the patient's ability to postpone treatment, advice should be sought from the attending physician.

in the case of antipsychotics and antiepileptics

For all parents:

* Presence of a history of neurological or neurodevelopmental disorders prior to the attacks except ADHD (epilepsy, head trauma with loss of consciousness of more than one hour, autism spectrum disorder autism spectrum disorder, intellectual disability, schizophrenia)
* Persons subject to a legal protection measure (safeguard of justice, curatorship, guardianship)
* Subject to a period of exclusion in the context of another research project
* Parent's refusal to participate in research

For parents carrying out the protocol on site:

* Person with contraindications to MRI
* For women of childbearing age, current or planned pregnancy
* Psychotropic products capable of modifying attention, vigilance and concentration taken less than 24 hours before questionnaires or examinations (sleeping pills and hypnotics, antipsychotics, mood regulators, antiepileptics and antihistamines). If in doubt about the patient's ability the patient's ability to postpone treatment, advice should be sought from the attending physician.

in the case of antipsychotics and antiepileptics

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Psychiatric nosography with MINI (parents) | During the one day of assessments
  Psychological interview
Assessment of PTSD symptoms severity in children 8-11 years and 12-17 years | During the one day of assessments
  Results from CPSS-5 a semi-structered interview
Assesssment of PTSD symptoms for parents and children over the age of 18 | During the one day of assessments
  Results from SCID-5-CV which is a semi-structered interview for the diagnosis of mental disorders DSM-5
Assessment of PTSD symptoms severity in adults | During the one day of assessments
  Scores from PCL-5 which is a self report measure
Secondary traumatisation | During the one day of assessments
  Parents and children : Scores from FST
Post-traumatic growth | During the one day of assessments
  Parents : Scores from PTGI
Coping skills for parents, children 12-17 years and over the age of 18 | During the one day of assessments
  Scores from BCI
Coping skills for parents and children 8-11 years | During the one day of assessments
  Scores from SRCS.
Resilience for parents and children over the age of 18 | During the one day of assessments
  Scores from ARM-R
Resilience for children 8 to 11 years old | During the one day of assessments
  Scores from CYRM-R-Child
Resilience for children 12 to 17 years old | During the one day of assessments
  Scores from CYRM-R-Youth
Attachment | During the one day of assessments
  Children : Scores from IPPA
Anxiety | During the one day of assessments
  Parents : scores from STAI
Depression | During the one day of assessments
  Parents : scores from BDI
Self-esteem | During the one day of assessments
  Parents : scores from SPP-Adult
Emotion regulation for parents and children over the age of 18 | During the one day of assessments
  Scores from ERQ
Emotion regulation for Children and adolescents aged 8 to 17 | During the one day of assessments
  Scores from ERQ-CA
Empathy for Parents, chidren 12-17 years and children over the age of 18 | During the one day of assessments
  Scores from BES-A
Empathy for Children 8-11 years | During the one day of assessments
  Scores from BES-C
World vision | During the one day of assessments
  Parents and children : scores from WAS
Well being | During the one day of assessments
  Parents and children : score from WHO-5
Assessment of Psychiatric nosography with CBCL/YSR (children) | During the one day of assessments
  Total score, Main scales: Internalized behaviours, Externalized behaviours, Subscales: Anxiety/Depression, Social withdrawal, Somatic complaints, Interpersonal problems, Thought disorder, Attention deficit disorder, Deviant behaviours, Aggressive behaviours, Other problems
Social support | During the one day of assessments
  Parents : scores from Social Support Questionnaire
Cognitive avoidance | During the one day of assessments
  Parents and children : scores from QEC
Bonding | During the one day of assessments
  Parents and children : scores from PBI
Familial functionning | During the one day of assessments
  Parents and children :Scores from the FAD-SF
Parenting style and practices | During the one day of assessments
  Parents and children : Scores from the APQ
Communication about 13-11 Event | During the one day of assessments
  Parents and children : results from Communication about 13-11 Event Interview
Attention | During the one day of assessments
  Parents and children : scores from the Attentional Network Test
Transmission of traumatic memory | During the one day of assessments
  Parents and children : results from the Approach-Avoidance Task
Executive functionning | During the one day of assessments
  Children : scores from BRIEF
Cortisol | During the morning of the one day of assessments
  Parents and children : Cortisol Awakening Response
Sleep - questionnaires for children 8-11 and 12-17 years | During the one day of assessments
  Scores from SDSC
Sleep - questionnaires for Parents and children over the age of 18 | During the one day of assessments
  Scores from PSQI
Sleep - questionnaires for Parents and children over the age of 18 | During the one day of assessments
  Scores from ISI
Sleep - actimetry Parents and children | One week before the one day of assessments
  Measurement of bedtimes and wake-up times using an actimeter (a wrist-worn watch-size device).
Sleep - planner Parents and children | One week before the one day of assessments
  Evalustion of the sleep diary
Neuroanatomical analysis | During the one day of assessments
  Parents and children : anatomic MRI with the classic anatomical sequences
Neurofunctional analysis | During the one day of assessments
  Parents and children fonctionnal MRI with the measurement of the magnitude of the BOLD signal

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère Guillery, Study Director — Université de Caen Normandie, Inserm, EPHE-PSL, PSL University, CHU de Caen, GIP Cyceron, U1077, NIMH, 14000 Caen, France
Locations (1):
- Umr-S 1077 Nimh, Caen, France

IPD SHARING:
Plan to Share IPD: No